CLINICAL TRIAL: NCT01053260
Title: Contingency Management for Promoting Weight Loss in University Students
Acronym: WeLCoMe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H09-067; 1R21HL092382-01A2 (NIH)
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Contingency Management; Weight Loss
Keywords: Contingency Management; Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LEARN Program (Active Comparator): Participants will receive weekly weight loss counseling based on the LEARN Program for Weight Management.
  Interventions: Behavioral: LEARN Program
- LEARN Plus Contingency Management (Experimental): Participants will receive weekly counseling based on the LEARN Program for Weight Management plus contingency management. Participants can earn chances to win prizes for losing weight and completing activities that promote weight loss.
  Interventions: Behavioral: LEARN Program; Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: LEARN Program — Participants will receive weekly counseling based on the LEARN Program for Weight Management
Behavioral: Contingency Management — Participants can earn chances to win prizes for losing weight and completing activities that promote weight loss.
  Arms: LEARN Plus Contingency Management

SUMMARY:
Rates of overweight and obesity are increasing, particularly among individuals aged 18 to 29. An estimated 25-35% of American college and university students are overweight or obese. Contingency Management (CM) is a behavioral intervention that provides tangible rewards for positive behaviors. CM has substantial evidence of efficacy in reducing smoking and drug use and increasing treatment retention and medication compliance. The current study will evaluate the efficacy of a 24-week CM intervention to promote weight loss in overweight and obese university students. Seventy participants with a body mass index (BMI) of 27.0-34.9 will be randomly assigned to one of two conditions: (a) LEARN, a manual guided behavioral weight loss program (Brownell, 2004), with weigh-ins and supportive counseling, or (b) LEARN with weigh-ins and supportive counseling plus CM. Participants in the CM condition will earn chances to win prizes each week in which they lose at least one pound. Once they lose 5% of baseline body weight, they will earn chances to win prizes for weight loss or weight maintenance. Additional chances can be earned by completing activities that promote weight loss. The primary outcomes will be absolute and proportional weight loss from pre- to post-treatment, as well as proportion of participants achieving clinically significant weight loss (>5% of baseline weight) and proportion moving into a lower risk BMI category. Secondary outcomes will include length of retention in the study, increase in physical activity level, and improvement in nutritional quality of diet. Effects of the CM intervention on psychiatric distress and self-efficacy and motivation to engage in activities that promote weight loss will also be assessed. We predict that participants in the CM condition will lose more weight than participants assigned to the LEARN program without CM, and that more CM participants will achieve clinically significant weight loss. We also predict that participants in the CM condition will remain in the program longer, show larger increases in physical activity, show greater improvements in diet quality, and have greater increases in levels of self-efficacy and motivation than comparison group participants. Mediators and moderators of CM outcomes will also be evaluated. If efficacious in promoting weight loss in a college population, CM could help to prevent or delay later development of obesity-related medical problems.

ELIGIBILITY:
Inclusion Criteria:

* currently enrolled as an undergraduate or graduate student
* age between 17 and 29 years
* body mass index in kg/m2 (BMI) between 27.0 and 39.9
* resting blood pressure between 90-140 (systolic) and 60-90 (diastolic) mmHg
* willingness and ability to participate for 24 weeks from date of enrollment
* willingness to be randomly assigned to one of two groups

Exclusion Criteria:

* serious acute or chronic medical problems (e.g. diabetes mellitus, heart disease, cancer, asthma, back or joint problems, hernias, history of recent surgery)
* pregnant or breast feeding
* current, uncontrolled psychiatric condition or serious psychiatric symptoms (e.g. current suicidality, psychotic symptoms
* meet criteria for a substance dependence disorder, (5) they report daily tobacco use
* any reported history of past or current eating disorders
* in recovery from pathological gambling
* report losing more than 10% of their heaviest body weight in the last 6 months
* report participation in a formal weight loss program in the last 6 months.

Ages: 17 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2010-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in Weight in Pounds | Baseline, 12 weeks, 24 weeks, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Petry, Ph.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States